CLINICAL TRIAL: NCT01232920
Title: First-line Antimetabolites as Steroid-sparing Treatment Uveitis Pilot Trial
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-00235
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Uveitis
Keywords: uveitis; antimetabolite; immunosuppressive; clinical trial
MeSH Terms: conditions — Uveitis | interventions — Methotrexate; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate
- Mycophenolate mofetil (Active Comparator)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Methotrexate — All methotrexate doses will be taken orally once per week in a divided dose (half in the morning, half in the evening), and should be taken with food. For the first two weeks, a loading dose of 15 mg/week orally will be administered to assess tolerability. After two weeks, the dose will be ramped up to 25 mg/week until the end of follow-up or until treatment failure due to intolerability, adverse events, or of lack of efficacy. If the study ophthalmologist decides to reduce the study treatment dose due to intolerability, the dose will be reduced to 20 mg per week while maintaining masking. If side effects persist and the study ophthalmologist wishes to reduce the dose a second time, the dose will be reduced to 15 mg per week.
  Arms: Methotrexate
Drug: Mycophenolate mofetil — Mycophenolate mofetil will be taken twice daily on an empty stomach. For the first two weeks, a loading dose of 500 mg/BID orally will be administered to assess tolerability. After two weeks, the dose will be ramped up to 1 g/BID until the end of follow-up or until treatment failure due to intolerability, adverse events, or lack of efficacy. If the study ophthalmologist decides to reduce the study treatment dose due to intolerability, the dose will be reduced to 750 mg/BID while maintaining masking. If side effects persist and the study ophthalmologist wishes to reduce the dose a second time, the dose will be reduced to 500 mg/BID.
  Other Names: Cellcept
  Arms: Mycophenolate mofetil

SUMMARY:
The proposed study is a masked trial, with stratified block randomization by site, designed to determine which treatment, methotrexate or mycophenolate mofetil, is more effective as first-line steroid-sparing treatment for patients with non-infectious uveitis requiring corticosteroid-sparing therapy.

One hundred non-infectious uveitis patients in need of corticosteroid-sparing therapy will be randomized to receive either oral methotrexate or oral mycophenolate mofetil at Aravind Eye Hospitals (Madurai and Coimbatore, South India). They will be followed monthly for 6 months after enrollment or until treatment failure. The investigators hypothesize that the proportion achieving corticosteroid-sparing success at 6 months for patients taking mycophenolate mofetil will be improved in comparison with patients taking methotrexate.

DETAILED DESCRIPTION:
Uveitis, a set of conditions defined by intraocular inflammation, is a significant cause of vision loss and morbidity in the United States and the world. The incidence was recently estimated to be more than 50 cases per 100,000 person-years, with a prevalence of approximately 115 per 100,000 persons. Additionally, uveitis is believed to be the cause of up to 10% of cases of legal blindness in the United States, or approximately 30,000 new cases of blindness per year. In contrast to common age-related eye disorders, uveitis may have a stronger socio-economic impact because it disproportionately affects younger working-age patients. Although the etiology of uveitis is varied, most cases are presumed to be immune-mediated and lack a known infectious cause. Even in developing countries such as India that have a larger burden of infection, the vast majority of cases are non-infectious.

The current mainstay of treatment for noninfectious uveitis is corticosteroids (topical, systemic, locally injected, or corticosteroid-eluting implants). Due to the well documented local and systemic side effects associated with corticosteroid therapy, other immunosuppressive therapies are frequently used as corticosteroid-sparing agents in patients who need long-term therapy. These include antimetabolites, calcineurin inhibitors, alkylating agents, and biologic drugs. Cost and morbidity associated with uncontrolled inflammation make the selection of an effective initial steroid-sparing agent extremely important.

It is common practice for patients requiring a steroid-sparing agent to be treated first with the less expensive methotrexate and then switched to mycophenolate mofetil in the event of treatment failure. However, results from non-comparative retrospective case series indicate that uveitis patients may be much more likely to achieve controlled inflammation and tolerate treatment with mycophenolate mofetil. Furthermore, approximately half of the patients who fail treatment with methotrexate go on to successful treatment with mycophenolate mofetil. There have been no prospective randomized, controlled trials to systematically determine which antimetabolite is more clinically efficacious as initial corticosteroid-sparing therapy, making it difficult for clinicians to make informed, evidence-based decisions about first-line immunosuppressive treatment.

Our contribution is expected to be a definitive understanding of the comparative efficacy, tolerability, and quality of life of these two antimetabolites as initial steroid-sparing therapy for uveitis patients requiring chronic therapy. This contribution is significant because it will enable clinicians to make evidence-based decisions when prescribing first-line immunosuppressive therapy for their uveitis patients. The use of optimal first-line therapy will improve quality of life by reducing the risk of vision loss and complications associated with uncontrolled ocular inflammation and long-term corticosteroid use.

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious anterior, intermediate, posterior or panuveitis
* Active uveitis within the last 60 days (defined by the presence of any of the following according to SUN criteria: ≥ 1+ anterior chamber cells, anterior vitreous cells, vitreous haze, active retinal or choroidal lesions)
* Prednisone dose ≥ 15 mg/day
* History of corticosteroid taper failure (inability to taper to prednisone 10 mg or less) or obvious chronic disease necessitating corticosteroid-sparing immunosuppressive treatment

Exclusion Criteria:

* Any infectious cause of uveitis
* Tuberculosis: Evidence of active TB (PPD and CXR required - latent TB patients are still eligible)
* Positive for Hepatitis: HBsAg and/or Hep C antibody
* Positive for Syphilis: RPR/VDRL and/or FTA-ABS
* Abnormal CBC (<2500 WBC or <75,000 Plts or <10 Hgb)
* Abnormal liver and/or kidney tests (ALT/AST >2x normal or CR>1.5)
* Pregnancy or breast-feeding (blood or urine pregnancy test for all females, excluding those who are post-menopausal)
* Chronic hypotony (IOP < 5 mm Hg for > 3 months)
* Prior use of any immunosuppressive drug for the treatment of uveitis in the past 6 months
* Prior failed treatment with methotrexate or mycophenolate mofetil
* Periocular or intravitreal corticosteroid injection in the past 3 months
* Fluocinolone acetonide implant surgery in either eye in < 3 years
* Intraocular surgery in < 30 days, or any ocular surgery scheduled during the 6-month study period
* VA of hand motions or worse in better eye
* < 16 years of age at enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S R Rathinam, MD, Principal Investigator — Aravind Eye Hospital; M B Babu, MD, Principal Investigator — Aravind Eye Hospital; Nisha Acharya, MD MS, Principal Investigator — Proctor Foundation, UCSF
Locations (2):
- India (2):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu

REFERENCES:
- [Derived] Niemeyer KM, Gonzales JA, Rathinam SR, Babu M, Thundikandy R, Kanakath A, Porco TC, Browne EN, Rao MM, Acharya NR. Quality-of-Life Outcomes From a Randomized Clinical Trial Comparing Antimetabolites for Intermediate, Posterior, and Panuveitis. Am J Ophthalmol. 2017 Jul;179:10-17. doi: 10.1016/j.ajo.2017.04.003. Epub 2017 Apr 14. PMID 28414043

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methotrexate | Mycophenolate Mofetil
Started | 41 | 39
Completed | 35 | 32
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (10.3) | 40.5 (14.2) | 40.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Treatment Success
Description: TREATMENT SUCCESS is defined as controlled ocular inflammation in both eyes with less than or equal to 10 mg/day of prednisone and/or 2 topical steroid drops/day sustained for 2 visits separated by at least 28 days (control of inflammation and prednisone dose must be achieved by 5-month visit and sustained until 6-month visit).
  Discontinuation of study medication at any time due to efficacy, tolerability, or safety may result in a declaration of TREATMENT FAILURE. Note that all patients will be classified as either a treatment success or failure.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 35 | 32
participants | 24 | 15
Statistical Analysis 1: Comparison: Methotrexate vs Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.09, Fisher Exact

2. Secondary Outcome: Time to Control of Inflammation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 35 | 32
days | 139 [62.5 to 142] | 124 [60 to 156]

3. Secondary Outcome: Change in Best Spectacle-corrected Visual Acuity (BSCVA)
Description: Change in best spectacle-corrected visual acuity (BSCVA) from baseline. Analysis on eye level
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 35 | 32
Number analyzed (Eyes) | 68 | 56
LogMAR | -0.26 (0.33) | -0.19 (0.36)

4. Secondary Outcome: Number of Eyes With Resolution of Macular Edema
Time Frame: 6 months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 35 | 32
Number analyzed (Eyes) | 68 | 56
Eyes
  Eyes with Macular Edema at Baseline | 22 | 13
  Eyes with Resolved Macular Edema | 17 | 7

ADVERSE EVENTS:
Arm/Group | Methotrexate | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/39
Other Adverse Events (participants affected / at risk) | 33/41 | 32/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=41) | Mycophenolate Mofetil (N=39)
Hospitalization (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin burn wound, not study related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=41) | Mycophenolate Mofetil (N=39)
Nausea (Gastrointestinal disorders) | 6 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 3 | 2
Systemic infection (Infections and infestations) | 3 | 4
Cataract (Eye disorders) | 5 | 3
Ocular hypertension (Eye disorders) | 4 | 2
Glaucoma (Eye disorders) | 2 | 2
Headache (General disorders) | 8 | 12
Fever for 12 hours (Infections and infestations) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No